CLINICAL TRIAL: NCT04744961
Title: Effect of Surgical Site Infections on Patient Reported Cosmetic Outcomes in Dermatologic Surgery
Status: Completed | Type: Observational
Sponsor: Region Skane (Other)
Responsible Party: Principal Investigator, Karim Saleh, Principal investigator, M.D, Ph.D, Region Skane
Other Study IDs: RegionSkane2021
Record Dates: First submitted 2021-02-03; First posted 2021-02-09 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Surgical Site Infection; Patient Satisfaction
MeSH Terms: conditions — Surgical Wound Infection; Patient Satisfaction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical site infections
  Interventions: Other: SCAR-Q survey
- Normal would healing
  Interventions: Other: SCAR-Q survey

INTERVENTIONS:
Other: SCAR-Q survey — Telephone survey

SUMMARY:
This study involves surveying two matched groups of patients that underwent dermatologic surgery at our department. One group had a documented surgical site infection and the other didn't. All patients will be asked to complete a questionnaire in which they assess the physical appearance of their scars and its psychosocial impact. Results will be compared between the groups.

DETAILED DESCRIPTION:
65 patients with a documented surgical site infection will be compared to 65 patients with normal wound healing in terms of patient reported outcome regarding scar physical appearance and psychosocial impact using SCAR-Q questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patient above 18 years of age that underwent a dermatosurgical procedure at our department between march 2017 and march 2020.

Exclusion Criteria:

* Patients assessed as not suitable for telephone survey due to hearing disabilities or cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All included patients had a surgical procedure performed at our department. One group had documented surgical site infections and the other didn't.
Sampling Method: Probability Sample
Enrollment: 114 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Comparing mean values of SCAR-Q scores in both groups | 3 months
  Scar-Q (http://qportfolio.org/scar-q/) is a patient reported outcome instrument in which scars will be assessed in terms of scar appearance and psychosocial impact. Scores will range from 0 (worst) to 100 (best). Scores will be compared between the two groups using either parametric or non-parametric tests depending on the distribution of the results.

SECONDARY OUTCOMES:
Association between patient characteristics and SCAR-Q scores | 3 months
  Score values (0-100) will be correlated to the following patient characteristics (gender, age, type of surgical procedure, anatomic location, and diagnosis of excised lesion)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of dermatology, Skåne university hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided